CLINICAL TRIAL: NCT03394456
Title: Technology to Improve the Health of Resource-poor Hispanics With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elizabeth Vaughan, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-40322; K23DK110341 (NIH); H-40322 (Other: Baylor College of Medicine IRB)
Record Dates: First submitted 2017-12-21; First posted 2018-01-09 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care; Community Health Workers

STUDY DESIGN:
Masking Description: In the last secondary study, there is single blinding (data collectors)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receive diabetes group visits/diabetes program
  Interventions: Other: diabetes program; Other: telehealth training and support for Community Health Workers
- Control (No Intervention): Receive usual care in the clinic, followed by group visits (wait list control) for cohorts 1-4 case-matched comparisons via chart review for cohort 5

INTERVENTIONS:
Other: diabetes program — Comprehensive diabetes program (weekly to bimonthly CHW mHealth contact (phone, text) for 12-months and monthly diabetes group visits for 6-months)
  Arms: Intervention
Other: telehealth training and support for Community Health Workers — weekly 1-hour diabetes training and patient support for CHWs via telehealth i.e., ZOOM technology for the study duration
  Arms: Intervention

SUMMARY:
This study evaluates the efficacy and implementation of a telehealth-supported, integrated diabetes group visit program led by Community Health Workers (CHWs). Primary study relates to efficacy and a secondary study addresses mentored implementation.

DETAILED DESCRIPTION:
The number of Hispanics diagnosed with diabetes is escalating in the US with disproportionately higher prevalence and complication rates than other ethnicities. CHWs are a well-established and culturally sensitive means to bridge gaps in care to individuals with diabetes. However CHWs are often left unsupported, placing patients at risk of substandard care or harm. Telehealth is a term used to describe a range of technologies to support healthcare delivery via communication with the patient or a member of the healthcare delivery team. Though telehealth has been implemented into diabetes programs for many years, there is a paucity of data showing the use of telemedicine for CHW training and support.

The primary study (n=89; Cohorts 1,2) compares clinical outcomes and treatment satisfaction of individuals who receive diabetes care in a 12-month telehealth supported, integrated CHW-led group visit program compared to those in usual care (wait list control). Group visits are 6-months and CHWs contact patients weekly to bimonthly (mobile health (mHealth)) for 12-months. This phase with have two cohort waves, separated by 6-months. The wait list control group for Cohort 2 will explore telehealth, clinician-patient encounters. A secondary study (n=59; Cohorts 3,4) at a new clinic evaluates the ability to implement the program. In the first phase of the secondary study the research team will conduct a RCT of individuals randomized to the diabetes program (intervention) vs usual care (control) to assess clinic feasibility. The clinic team will observe this process and learn the project protocols during Phase 1. In the second phase, the clinic team will lead the group visits while the research team mentors them to conduct the project in-person at the group visits and via telehealth each week (ZOOM video conferencing). Another secondary study (n=138; Cohort 5) aims to expand the reach of the education and CHW intervention for individuals who may not be able to or cannot come to the clinic for group visits. Specifically, individuals will received the education from the program monthly via a secure text message video, CHWs will contact weekly to bimonthly to advocate for their needs, and participants will receive their routine care as usual in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic adults with diabetes, low-income (earn less than/equal to 250% federal poverty level)

Exclusion Criteria:

* not able to understand Spanish, group visit is not appropriate for care i.e., need individualized care, pregnancy, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-01-13 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Glycemic control | At baseline and every 6-months until study completion
  Hemoglobin A1c (%)

SECONDARY OUTCOMES:
Adherence to preventive care guidelines | pre/post diabetes group visits
  As measured by placement on a statin, annual urine micro albumin, target A1c, weight loss (if applicable), retinal eye examination, blood pressure targets, serum B12 measurements, vaccinations.
Survey | at the beginning and end of each cohort (baseline, six-months)
  The survey totaled 12 questions and assessed participant satisfaction, mental relaxation, faith/spirituality, and open-ended comments. Questions were ranked as followed: 1-3 (4-point Likert Scale), 4-7 (10-point Likert Scale), 8-11 (open-ended, descriptive), 12 (days of exercise/week). The Use of Mental Stress Management/Relaxation Techniques questionnaire and our pilot study survey templates were used to evaluate patient group visit and CHW satisfaction. We defined acceptability as high (3.5-4/4 or 8-10/10), moderate (2-3.4/4 or 4-7/10), and low (1-1.9/4 or 1-3/10) and totaled the items to create an overall score.
Diabetes-related health | at the beginning and end of each cohort (baseline, six-months)
  As measured by the Self Management Resource Center Surveys: Diabetes Medications (a 4-question yes/no survey to assess patient medication adherence and understanding of their medications), Self-rated Health (a 1-question ranked on a 5-point scale (1 is excellent, 5 is poor) to determine the patient's view of their health)
Body Mass Index (BMI) | At baseline and every 6-month until study completion
  Body Mass Index (BMI) (weight in kg/height in m^2)
Blood Pressure | At baseline and every 6-month until study completion
  Blood Pressure (mmHg)
Barriers to care | weekly to bimonthly from baseline to 12-months
  We obtain barriers to care data from the CHW-patient mobile health (mHealth) records and chart review, and group into three categories: obtaining medications, appointment access, clinic eligibility. mHealth records were sent to the study physician through a secure, encrypted site on a weekly basis.
longitudinal outcomes | from the time group visits end and as long as month-24 after
  conduct a chart review to determine long-term (until 24-months post group visits) clinical outcomes including blood pressure (mmHg)
longitudinal outcomes | from the time group visits end and as long as month-24 after
  conduct a chart review to determine long-term (until 24-months post group visits) clinical outcomes including HbA1c (%)
longitudinal outcomes | from the time group visits end and as long as month-24 after
  conduct a chart review to determine long-term (until 24-months post group visits) clinical outcomes including BMI (kg/m^2)

OTHER OUTCOMES:
Feasibility and acceptability of telehealth patient, clinician encounters during diabetes group visits | At six months after group visits for wait list control Cohort 2
  As measured by the Telehealth Usability Questionnaire(21-question survey where 1 is strongly disagree and 5 is strongly agree)
Feasibility and acceptability of telehealth support for community health workers 2 | At baseline and six months during Cohort 1 intervention group
  The Diabetes Knowledge Test (University of Michigan, 2015; 23 questions; where a total score of 0 indicates the least and 23 indicates the most diabetes knowledge based on this test)
Feasibility and acceptability of telemedicine support for community health workers | After each cohort (every six months)
  As measured by a six-month 4-question survey (four open-ended questions i.e., what CHWs liked, disliked, general comments) and a 10-question multiple choice posttest that covers content they were taught the last six months (Vaughan et al, 2018)
Feasibility and acceptability of telemedicine support for community health workers | After Cohort 1
  As measured by the Telehealth Usability Questionnaire(21-question survey where 1 is strongly disagree and 5 is strongly agree)
CHW knowledge | During Cohort 2 at baseline (TEST-1 pretest), 6- (TEST-1 posttest, TEST-2 pretest) and 12-months (TEST-2 posttest)
  As measured by pre- /post-tests. TEST-1 (n=21 questions) and TEST-2 (n=19 questions). Tests were multiple choice with 3-5 answer option and were original to this study.
CHW knowledge | During the secondary study, at baseline and 6-months (pre/posttest)
  This will be accomplished by the 24-question Starr County Diabetes Knowledge Test, which has shown validity and reliability in English and Spanish. Each of the 24-question has three answer choices. This will be pre/posttest format.
Access to care | from baseline to 12-months
  As measured by the amount of contact participants had with the clinic during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Vaughan, DO, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peek ME, Cargill A, Huang ES. Diabetes health disparities: a systematic review of health care interventions. Med Care Res Rev. 2007 Oct;64(5 Suppl):101S-56S. doi: 10.1177/1077558707305409. PMID 17881626
- [Background] Dias S, Gama A. [Community-based participatory research in public health: potentials and challenges]. Rev Panam Salud Publica. 2014 Feb;35(2):150-4. Portuguese. PMID 24781097
- [Background] Mbuagbaw L, Thabane L, Ongolo-Zogo P, Lang T. The challenges and opportunities of conducting a clinical trial in a low resource setting: the case of the Cameroon mobile phone SMS (CAMPS) trial, an investigator initiated trial. Trials. 2011 Jun 9;12:145. doi: 10.1186/1745-6215-12-145. PMID 21658262
- [Background] Furino A. ￼Community Health Worker National Workforce Study. Wasthington, DC: US Dept of Health and Human Services; 2007.
- [Background] Norris SL, Chowdhury FM, Van Le K, Horsley T, Brownstein JN, Zhang X, Jack L Jr, Satterfield DW. Effectiveness of community health workers in the care of persons with diabetes. Diabet Med. 2006 May;23(5):544-56. doi: 10.1111/j.1464-5491.2006.01845.x. PMID 16681564
- [Background] Lujan J, Ostwald SK, Ortiz M. Promotora diabetes intervention for Mexican Americans. Diabetes Educ. 2007 Jul-Aug;33(4):660-70. doi: 10.1177/0145721707304080. PMID 17684167
- [Derived] Vaughan EM, Virani S, Al Rifai M, Cardenas VJ Jr, Johnston CA, Porterfield L, Santiago Delgado Z, Samson SL, Schick V, Naik AD. Determining call-to-entry rate and recruitment barriers in clinical studies for community clinics serving low-income populations: a cohort study. BMJ Open. 2023 Oct 28;13(10):e077819. doi: 10.1136/bmjopen-2023-077819. PMID 37898484
- [Derived] Vaughan EM, Cardenas VJ Jr, Chan W, Amspoker AB, Johnston CA, Virani SS, Ballantyne CM, Naik AD. Implementation and Evaluation of a mHealth-Based Community Health Worker Feedback Loop for Hispanics with and at Risk for Diabetes. J Gen Intern Med. 2024 Feb;39(2):229-238. doi: 10.1007/s11606-023-08434-7. Epub 2023 Oct 6. PMID 37803098
- [Derived] Vaughan EM, Hyman DJ, Naik AD, Samson SL, Razjouyan J, Foreyt JP. A Telehealth-supported, Integrated care with CHWs, and MEdication-access (TIME) Program for Diabetes Improves HbA1c: a Randomized Clinical Trial. J Gen Intern Med. 2021 Feb;36(2):455-463. doi: 10.1007/s11606-020-06017-4. Epub 2020 Jul 22. PMID 32700217

DOCUMENTS (1):
  • Informed Consent Form (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT03394456/ICF_000.pdf